CLINICAL TRIAL: NCT00604747
Title: The Effects of Practice Structure on Motor Learning in Post-Stroke Patients
Brief Title: Practice Structure on Motor Learning in Post-Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Camila Torriani, University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0038.0.254.000-05; 0038.0.254.000-05
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2008-01-30 (Estimated); Status verified 2008-01

CONDITIONS: Stroke
Keywords: motor learning; hemiplegia; stroke; practice; physiotherapy
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1, 2 (Other)
  Interventions: Other: Structure practice

INTERVENTIONS:
Other: Structure practice — there were 2 groups which received random practice and constant practice during acquisition phase
  Other Names: experimental group (EG); control group (CG)

SUMMARY:
Background: The literature indicates that, in relation to motor learning, healthy subjects benefit more from random practice than from constant practice. However, this effect is not well known in post-stroke patients. Objective: The goal of this study was to investigate the effects of practice structure on motor learning in post-stroke patients. Methods: Participants included an experimental group (EG) of post-stroke patients: 17 males and females; and a control group (CG) of healthy individuals: 17 males and females. At the acquisition phase, all participants performed 30 trials of a coincident timing task. Nine individuals from each group practiced constantly (C) at a stimulus propagation speed of 3 mph, and eight from each group practiced randomly (R) at speeds of 2, 3, and 5 mph. Subsequent phases included: 1) transfer, 2) retention after 15 minutes, and 3) retention after 3 days. Each of these phases included 20 trials: 10 at a speed of 1 mph, and 10 at a speed of 4 mph. Intra- and inter-group comparisons were made employing an alpha level of 0.05 (5%).

DETAILED DESCRIPTION:
Utilized was Bassin's anticipation timer (Lafayette Instruments #50575), which is comprised of a control screen, one 1.52 m gutter with 32 diodes placed on it linearly, and a response button. The screen has a digital display, with commands that permit the operator to control the stimulus propagation speed and the preparatory interval speed. Once activated, the screen exhibits an alert signal, and, after the preparatory interval, it initiates the propagation of a luminous stimulus, lighting the 32 diodes successively. The task required participants to press the response button simultaneously with the illumination of the last diode. The digital display showed the error measure (em): that is, the difference between the illumination of the last diode and the response.

ELIGIBILITY:
Inclusion Criteria:

1. First cerebrovascular accident
2. Lesion covering the middle and the anterior cerebral artery territories
3. Presence of hemiplegia or hemiparesis
4. Mini-Mental State Examination (MMSE) score above 24 (19)
5. Sufficient attention and comprehension to perform the task
6. Absence of other associated neurological diseases.

Exclusion Criteria:

1. Acute medical problems
2. Uncorrected vision loss
3. Previous history of psychiatric admission
4. History of multiple strokes, transient ischemic attacks
5. Pathology of the less affected, ipsilateral to stroke upper extremity that would affect ability to perform the task
6. Score of 23 or less on the MMSE
7. Difficulty in comprehension of verbal command and simple instructions
8. Aphasia of comprehension.

Ages: 40 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2006-08; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
change in performance during the acquisition; performance exhibited during the transfer phase was maintained during retention phases 1 and 2; and differences between the groups during the transfer phase and retention phases | time in miliseconds

CONTACTS AND LOCATIONS:
Overall Officials: Camila Torriani, Principal Investigator — University of Sao Paulo; Camila Torriani, Study Chair — University of Sao Paulo
Locations (1):
- Camila Torriani, São Paulo, São Paulo, Brazil